CLINICAL TRIAL: NCT00003407
Title: Treatment of Poor Prognosis Acute Myeloid Leukemia and Blastic Crisis Chronic Myelogenous Leukemia With Mylotarg, High-Dose Cytarabine, Mitozantrone and Ethyol AML/CML 2000-06.
Brief Title: Amifostine & High-Dose Combination Chemotherapy in Treating Patients With Acute ML or CML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The P.I deceased.
Sponsor: Rush University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000066416; P01CA075606 (NIH); ALZA-RUSH-AML-9801 (Registry Identifier: ALZA); NCI-V98-1447 (Other Grant/Funding Number: NCI); RUSH-AML-9801 (Other: Rush University Medical Center)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia; Myelodysplastic Syndromes; Neutropenia
Keywords: recurrent adult acute myeloid leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute myeloid leukemia; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; drug/agent toxicity by tissue/organ; neutropenia
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Myelodysplastic Syndromes; Neutropenia; Leukemia, Myeloid, Acute; Blast Crisis | interventions — Amifostine; Cytarabine; Mitoxantrone

ARMS (1):
- Effectiveness of amifostine &high-dose combination chemotherapy in treating patients with AML or CML (Experimental): Treatment of Newly Diagnosed High Risk And Relapsed Acute Myeloid Leukemia and Blastic Crisis Chronic Myelogenous Leukemia With Ethyol and High-Dose Cytarabine + Mitoxantroni, followed by Maintenance Phase Using Low-Dose ARA-C, rhGM-CSF, Pentoxifylline, Ciprofloxacin, and Decadron
  Interventions: Drug: amifostine trihydrate; Drug: cytarabine; Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cytarabine
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of amifostine and high-dose combination chemotherapy in treating patients with acute myeloid leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the effects of amifostine on the response to remission induction therapy and consolidation with cytarabine and mitoxantrone in patients with poor prognosis acute myeloid leukemia (AML), relapsed AML, and blastic phase chronic myelogenous leukemia (CML). II. Assess the effects of amifostine on the biology of AML and CML cells in vivo in this patient population.

OUTLINE: Patients receive treatment prior to induction therapy on protocols CYL 90-03 and CYL 97-59. Induction therapy consists of amifostine IV on days 1 and 5 and three times a week from days 6 to 28. Fifteen minutes after amifostine on days 1 and 5, patients receive cytarabine IV over 3 hours at hour 0 and hour 12 and mitoxantrone IV over 1 hour at hour 15. Patients who do not enter remission receive a second course of induction therapy. Patients with persistent AML following a second course are removed from the study. Patients who achieve a complete response (CR), clinical CR, or remission in bone marrow but without hematologic recovery or who return to myelodysplastic syndrome receive consolidation therapy. Consolidation therapy consists of amifostine IV on days 1 and 5 and then three times a week until blood counts recover or day 30, whichever comes first. Patients also receive cytarabine and mitoxantrone as in induction therapy. Patients receive a second course of consolidation therapy beginning 1 week after blood counts recover. After completion of consolidation therapy, patients are enrolled on protocol MDS 97-53.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* DISEASE CHARACTERISTICS: Newly diagnosed high-risk acute myeloid leukemia (AML) defined as AML after myelodysplastic syndrome; refractory anemia with excess blasts in transformation or "AML in evolution" also eligible AML following a chronic myeloproliferative disorder (except chronic myelogenous leukemia).
* Therapy-related AML or AML following exposure to a known hematopoietic toxin Relapsed AML Age 70 or older OR AML in first relapse defined as
* AML in first relapse without treatment on protocol AML-9801 Relapsed following standard chemotherapy Previously treated on AML-9701 and relapsed after at least 6 months of remission OR Chronic myelogenous leukemia (CML) in blast crisis defined as
* 20% or more blast cells in the bone marrow or peripheral blood Pure lymphoid blastic crisis eligible if resistant to an acute lymphocytic leukemia type treatment regimen or relapsed after initial response to such treatment.
* PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy
* Not specified Hematopoietic:
* Not specified Hepatic: Bilirubin less than 3 mg/dL SGOT/SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine less than 3 mg/dL Cardiovascular:
* No overt congestive heart failure or uncontrollable ventricular arrhythmias
* No uncontrollable hypertension Neurologic: No cerebellar dysfunction
* Other Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception.
* PRIOR CONCURRENT THERAPY: See Disease Characteristics above.

Exclusion criteria:

-Not identified by the protocol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-02-13 (Actual); Primary Completion 2004-04-07 (Actual); Study Completion 2004-04-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of amifostine and high-dose combination chemotherapy in treating patients with acute myeloid leukemia or chronic myelogenous leukemia | 6 months
  Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Philip D. Bonomi, MD, Study Chair — Rush University Medical Center
Locations (4):
- United States (4):
  - Cook County Hospital, Chicago, Illinois
  - Rush Cancer Institute, Chicago, Illinois
  - Angelo P. Creticos, M.D. Cancer Center, Chicago, Illinois
  - Rush-Riverside Cancer Center, Kankakee, Illinois

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/search/results?swKeyword=RUSH-AML-9801